CLINICAL TRIAL: NCT05471050
Title: The Combination of Tacrolimus and Danazol as the Treatment of Steroid-resistant/Relapse Immune Thrombocytopenia: A Randomized, Controlled, Open-label Trial
Brief Title: The Combination of Tacrolimus and Danazol as the Treatment of Steroid-resistant/Relapse Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-ITP036
Record Dates: First submitted 2022-07-17; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Immune Thrombocytopenia
Keywords: Immune Thrombocytopenia; tacrolimus; danazol
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Danazol

STUDY DESIGN:
Intervention Model Description: The investigators are undertaking a randomized controlled trial of 120 adults with steroid-resistant/ relapse ITP in China. Patients were randomized to tacrolimus plus danazol and danazol monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tacrolimus and Danazol (Experimental): Tacrolimus is given at a dose of 0.03mg/kg·d, and the dose is adjusted to maintain the trough concentration of tacrolimus at approximately 3-5 ng/mL for 12 weeks.
  Interventions: Drug: TAC; Drug: Danazol
- Danazol (Active Comparator): Danazol is given at 200mg bid for 12 weeks.
  Interventions: Drug: Danazol

INTERVENTIONS:
Drug: TAC — Tacrolimus is given at a dose of 0.03mg/kg·d, and the dose is adjusted to maintain the trough concentration of tacrolimus at approximately 3-5 ng/mL for 12 weeks.
  Arms: tacrolimus and Danazol
Drug: Danazol — Danazol is given at 200mg bid for 12 weeks.

SUMMARY:
Randomized, open-label, multicenter study to compare the efficacy and safety of combination of tacrolimus and danazol versus danazol for the treatment of adults with steroid-resistant/relapse immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a randomized controlled trial of 120 adults with steroid-resistant/relapse ITP in China. Patients were randomized to tacrolimus plus danazol and danazol monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Primary immune thrombocytopenia (ITP);
* 18 years older;
* Platelet count of less than 30×10^9/L at enrollment;
* Patients who did not achieve a sustained response to treatment with full-dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid-tapering or after its discontinuation;
* Patients who were receiving other maintenance regimens, primarily corticosteroids, ciclosporin, or mycophenolate mofetil, were also eligible if the dose of treatment had been stable in the past month and the dose was expected to be stable after enrolment and remained unchanged at least for the first 4 weeks of study until initial response was assessed, unless severe adverse events were suspected.

Exclusion Criteria:

* Secondary ITP (e.g., patients with HIV, HBV, HCV, Helicobacter pylori infection or SLE);
* Congestive heart failure, severe arrhythmia;
* Nursing or pregnant women;
* ALT or AST levels ≥ 3× the upper limit of the normal threshold;
* Creatinine or serum bilirubin levels ≥ 1.5× the upper limit;
* Active or previous malignancy ;
* Patients who had received danazol treatment or did not respond to danazol;
* Patients unable to have routine blood tests because of reasons such as insufficient time.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Sustained response | 6 months
  Sustained response was defines as the maintenance of platelet count ≥ 30 x 10^9/L, and at least 2-fold increase of the baseline count, and the absence of bleeding, and no need for rescue medication at the 6-month follow-up.

SECONDARY OUTCOMES:
Complete response | 6 months
  Complete response was defines as the maintenance of platelet count ≥ 100 x 10^9/L, and at least 2-fold increase of the baseline count, and the absence of bleeding, and no need for rescue medication.
Response | 6 months
  Response was defines as the maintenance of platelet count ≥ 30 x 10^9/L, and at least 2-fold increase of the baseline count, and the absence of bleeding, and no need for rescue medication.
Time to response | 6 months
  Time to response was defined as the time from starting treatment to the time to achieve the response.
Duration of response | 6 months
  Duration of response was measured from the achievement of response to the loss of response.
Adverse events | 6 months
  Adverse events were scaled according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — Peking University People's Hospital, Peking University Insititute of Hematology
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China